CLINICAL TRIAL: NCT06939296
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of VCT220 Tablets in Overweight or Obese Participants
Brief Title: A Research Study of VCT220 in Adult Chinese Participants With Obesity
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vincentage Pharma Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VCT220-III-01
Record Dates: First submitted 2025-04-10; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- High dose group (Experimental): Participants will receive VCT220 orally, once daily, titrate during 8 weeks and maintain at a high dose.
  Interventions: Drug: VCT220
- Moderate dose group (Experimental): Participants will receive VCT220 orally, once daily, titrate during 6 weeks and maintain at a moderate dose.
  Interventions: Drug: VCT220
- Placebo group (Placebo Comparator): Participants will receive placebo tablets orally, once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VCT220 — A small molecule GLP-1R drug, film coated tablet
  Other Names: CX11
  Arms: High dose group; Moderate dose group
Drug: Placebo — Placebo tablets
  Arms: Placebo group

SUMMARY:
The main purpose of this study is to assess how VCT220 tablets affect the bodyweight in obese or overweight adult participants. Participant will be randomly assigned to the high-dose group, low-dose group, or placebo group. Each participant will take the study drug orally once daily for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years, both male and female;
* At screening, BMI ≥ 28 kg/m² or 24 kg/m² ≤ BMI < 28 kg/m² with at least one of the following conditions:

  1. Comorbid prediabetes (impaired fasting glucose and/or abnormal glucose tolerance), hypertension, dyslipidemia, or fatty liver (within the past 6 months prior to screening);
  2. Comorbid weight-bearing joint pain (as determined by the investigator, excluding joint pain caused by other diseases);
  3. Obesity-related shortness of breath or obstructive sleep apnea syndrome;
* Weight change during the past 3 months due to diet and exercise control should not exceed 5% (self-reported); weight change calculation formula: (highest weight - lowest weight in the past 3 months) / highest weight * 100%;
* Willing and able to maintain a stable diet and exercise regimen throughout the study;
* Fully understands the purpose of the study, able to communicate well with the investigator, can comprehend and comply with the requirements of this study, and is willing to sign the informed consent form

Exclusion Criteria:

* Patients with type 1, type 2, or other types of diabetes.
* A history of endocrine diseases or obesity caused by single gene mutations, including but not limited to hypothalamic obesity, pituitary obesity, hypothyroid obesity, Cushing's syndrome, insulinoma, acromegaly, and hypogonadism.
* A history of weight-loss surgery (except for liposuction performed more than 1 year ago) or plans to undergo weight-loss surgery, use weight-loss devices, or medical equipment during the study.
* Has used any of the following medications or treatments:

  1. Has previously used any GLP-1 receptor agonists (GLP-1RAs), GLP-1-related multi-target agonists (such as GLP-1/glucose-dependent insulinotropic peptide [GIP] dual receptor agonists, GLP-1 receptor/glucagon receptor [GCGR] dual agonists, GLP-1/GIP/glucagon [GCG] triple receptor agonists, etc.), or combination formulations containing GLP-1RAs (such as exenatide, liraglutide, semaglutide, benaglutide, etc.);
  2. Within the past 6 months prior to screening, has used any approved or unapproved weight-loss medications other than GLP-1 receptor agonists (GLP-1RAs) and GLP-1-related multi-target agonists (such as orlistat, phentermine/topiramate, naltrexone/bupropion, etc.), or weight-affecting herbal medicines, supplements, meal replacements, etc.;
  3. Within the past 3 months prior to screening, has used any antidiabetic medications, such as metformin, α-glucosidase inhibitors, sulfonylureas, dipeptidyl peptidase-4 (DPP-4) inhibitors, sodium-glucose co-transporter-2 (SGLT-2) inhibitors, thiazolidinediones (TZDs), etc.;
  4. Within the past 3 months prior to screening, has used any medications that may cause significant weight gain, including systemic corticosteroid treatment for more than 1 week, tricyclic antidepressants, antipsychotic or anticonvulsant medications (e.g., imipramine, amitriptyline, mirtazapine, paroxetine, phenelzine, chlorpromazine, clozapine, olanzapine, valproic acid and its derivatives, lithium salts, methyldopa, etc.).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Actual)
Dates: Start 2024-12-24 (Actual); Primary Completion 2025-10-25 (Estimated); Study Completion 2026-03-27 (Estimated)

PRIMARY OUTCOMES:
Percentage change from baseline in body weight | From baseline to week 34
The proportion of subjects with a body weight reduction ≥5% from baseline | From baseline to week 34

SECONDARY OUTCOMES:
Percentage change from baseline in waist circumference | From baseline to week 34
Percentage change from baseline in body weight | From baseline to week 52
The proportion of subjects with a body weight reduction of ≥10%, ≥15%, and ≥20% | From baseline to week 34 and week 52
The proportion of subjects with a body weight reduction of ≥5% from baseline | From baseline to week 52
Percentage change from baseline in body mass index (BMI) | From baseline to week 52
Percentage change from baseline in waist circumference | From baseline to week 52
Percentage change from baseline in blood pressure | From baseline to week 52
  DBP and SBP
Percentage change from baseline in blood lipid profiles | From baseline to week 52
  TC, TG, LDL-C, and HDL-C
Percentage change from baseline in fasting plasma glucose | From baseline to week 52
Percentage change from baseline in fasting insulin | From baseline to week 52
Percentage change from baseline in Glycosylated Hemoglobin (HbA1c) | From baseline to week 52
Improvement in quality of life | From baseline to week 52
  Measured by Impact of Weight on Quality of Life-Lite Clinical Trials questionnaire（IWQoL-Lite-CT ). The IWQoL-Lite-CT has 20 items, each scored on a 5-point Likert scale, with a total score of 100. Higher scores indicate less negative impact of weight on quality of life.
Improvement in quality of life | From baseline to week 52
  Measured by Medical Outcomes Study 36-Item Short-Form Health Survey questionnaire version 2 (SF-36 v2) . It contains 36 items grouped into 8 domains, Each item is scored based on a predefined scale. Higher scores indicate better health-related quality of life.

OTHER OUTCOMES:
Adverse events, including treatment-emergent adverse events (TEAEs), serious adverse events (SAEs) | From week 0 to week 56
Change from baseline in liver fat content measured by Magnetic Resonance Imaging Proton Density Fat Fraction (MRI-PDFF) | From baseline to week 52

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital （ There are multiple sites in this clinical trial）, Beijing, Beijing Municipality, China